CLINICAL TRIAL: NCT03638895
Title: Randomised Controlled Trial to Evaluate Impact of Energy Expenditure Information on the Outcome of Weight Loss During a Standardised Multicomponent Weight Management Intervention
Brief Title: Energy Expenditure From ECAL Indirect Calorimeter in a Multicomponent Weight Management Service
Acronym: ECAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Metabolic Health Solutions UK (Unknown)
Responsible Party: Principal Investigator, Prof. John Wilding, Professor of Medicine & Honorary Consultant Physician, Obesity and Endocrinology Research, Theme Lead for Metabolism and Nutrition, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UoL001379
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Severe Obesity; Sleep Apnoea
Keywords: weight management; obesity; severe obesity; structured dietary intervention; calorie restriction; indirect calorimetry; resting energy expenditure; resting metabolic rate; respiratory quotient; substrate oxidation; glycemic variability; insulin sensitivity; peripheral neuropathy
MeSH Terms: conditions — Obesity; Obesity, Morbid; Sleep Apnea Syndromes; Insulin Resistance; Peripheral Nervous System Diseases | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Practitioner) Energy expenditure information (resting energy expenditure & respiratory quotient) is withheld from participant and practitioner providing care to participants in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECAL group (Active Comparator): Intervention group (ECAL) - practitioners and participants receive measured energy information from ECAL indirect calorimeter including resting energy expenditure and respiratory quotient to diagnose, manage and advise on modification of caloric restriction and physical activity level. Energy information also allows participant and practitioner to monitor and compare changes to their metabolic health throughout the duration of intervention.
  Interventions: Device: ECAL Indirect Calorimeter
- SC group (Placebo Comparator): Standard care (SC) - participants receive standard care (diet, exercise & behaviour modification therapy) as part of the multicomponent weight management intervention within the tier 3 weight management service. Practitioners will rely on standard predictive equations to provide dietary advice and intervention.
  Interventions: Behavioral: Diet, exercise & behaviour modification therapy

INTERVENTIONS:
Device: ECAL Indirect Calorimeter — The ECAL is an open-circuit portable indirect calorimeter that measures both volume of CO2 expired and O2 consumed using a small mixing chamber. Participants will breathe through a mouthpiece with a nose clip applied whilst lying in a restful and comfortable position for 15 minutes. ECAL device will provide breath-by-breath measurements of the resting energy expenditure and respiratory quotient which will allow both practitioners and participants to monitor their metabolic health and compare the effect of dietary and physical activity intervention over the course of the structured intensive lifestyle intervention (24-weeks).
  Arms: ECAL group
Behavioral: Diet, exercise & behaviour modification therapy — Standard care (SC) - participants receive standard care (diet, exercise & behaviour modification therapy) as part of the multicomponent weight management intervention within the tier 3 weight management service. Practitioners will rely on standard predictive equations to provide dietary advice and intervention.
  Arms: SC group

SUMMARY:
Whether greater weight loss is as a result of a smaller reduction in energy expenditure with caloric restriction is not known. Resting energy expenditure and 24-hour energy expenditure vary substantially between individuals. In some cases, relatively reduced rates of 24h EE predict weight gain in some populations who have high prevalence of obesity. Obese individuals that lose weight experience a decrease in 24-h EE and resting energy expenditure that is lower than predicted based on changes in body composition. Most weight loss studies have found a large individual variation in the amount of weight change, and whether an individual's response to an intervention can be predicted is not clear. Measurements of 24-hour EE in response to fasting may help predict weight loss. The ECAL indirect calorimeter (ECAL) is a validated device purpose-built to provide the practitioner and patient with energy information that allows for more accurate, reliable method of establishing an obese individuals' metabolic profile. The aim of this study is to determine whether providing energy information from ECAL indirect calorimeter as an adjunct to the multicomponent weight management intervention in non-diabetic obese and severely obese individuals would help predict the response of weight loss.

DETAILED DESCRIPTION:
Weight loss is important to improve overall health and reduce risk of obesity-related comorbidities such as diabetes. Numerous studies performed on individuals with predisposed genetic propensity to obesity who are deemed to be metabolically 'thrifty', require further structured intensification of caloric restriction and change in physical activity in order to achieve weight loss. Whether greater weight loss is as a result of smaller reduction in energy expenditure with calorie restriction is not known. Resting energy expenditure and 24-hour energy expenditure vary substantially between individuals. Obese individuals that lose weight experience a decrease in 24-h EE and resting energy expenditure that is lower than predicted based on changes in body composition. Most weight loss studies have found a large individual variation in the amount of weight change, and whether an individual's response to an intervention can be predicted is not clear. Measurements of 24-hour EE in response to fasting may help predict weight loss. The ECAL indirect calorimeter (ECAL) is a validated device purpose-built to provide the practitioner and patient with energy information that allows for more accurate, reliable method of establishing an obese individuals' metabolic profile. The ECAL device also measures the respiratory quotient (RQ) which is the ratio of the volume of carbon dioxide expired to that of oxygen consumed by the individual for every breath. Previous studies demonstrated variability in role of RQ in predicting weight loss, but individuals who demonstrated an RQ in the lower range (<0.72) were more likely to maintain the weight-loss achieved on a caloric restriction and avoid a weight loss rebound as compared to those with RQ in the higher range (>0.75). This suggests that RQ could prove useful in clinical practice as a prognostic marker for long-term effectiveness of low- and very-low-calorie diets used to induce weight loss. Baltimore Longitudinal Study on Aging shared a similar finding that fasting RQ or respiratory exchange ratio adjusted for age, BMI, and fat free mass was positively related to weight change. The aim of this study is to determine whether providing energy information from ECAL indirect calorimeter as an adjunct to the multicomponent weight management intervention in non-diabetic obese and severely obese individuals would help predict the response of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI > or equivalent to 30 kg/m2 to - 60 kg/m2
* Stable weight (change of <5% within 12 weeks before screening based on medical history)
* Subjects are well-motivated, capable and willing to learn how to undergo indirect calorimetry testing
* Willing and able to adhere to prohibitions and restrictions specified within this protocol

For Subjects participating in the glycaemic variability sub-study:

* Subject understands instructions on the use of continuous glucose monitor sensor and is willing to undergo appropriate training and testing

Exclusion Criteria:

* Taking weight loss medication within 12 weeks prior to randomisation
* Previous or planned bariatric surgery
* History of Type 1, Type 2 diabetes mellitus, DKA or diabetes secondary to pancreatitis
* Has HbA1c > or equal to 6.5% or Fasting Plasma Glucose > or equal to 7.0 mmol/L at screening.

NOTE: a one-time repeat measurement is allowed, if value of HbA1c and/or FPG is not consistent with prior values

* History of obesity with a known secondary cause (Cushing's disease/syndrome)
* Oral corticosteroid use (except in the short term use of a 7-10 day course)
* Ongoing, inadequately controlled thyroid disorder defined as thyroid-stimulating hormone > 6 mIU/litre or < 0.4 mIU/litre
* History of malignancy within 3 years before screening (or diagnosis of malignancy within this period)
* estimated glomerular filtration rate < 30 ml/min/1.73m2 on serum testing
* Alanine aminotransferase level is <2.0 times the upper limit of normal or total bilirubin is >1.5 times the upper limit of normal at screening
* Other major illness likely to preclude participation in the trial
* History of glucagonoma
* A myocardial infarction, unstable angina, revascularisation procedure (stent or bypass graft surgery) or cerebrovascular accident within 12 weeks before screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Magnitude of weight loss (in kg) | 6 months

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | 6 months
  The measurement of number of calories that the body burns at rest in 24 hours, expressed as kcal/day
Respiratory Quotient (RQ) | 6 months
  The ratio of carbon dioxide production to oxygen consumption and reflects the relative contribution of fat, carbohydrate, and protein in the oxidation fuel mixture.
Secretion of gut hormones (GLP-1, GIP, PYY) | 6 months
  Secretion of appetite regulating gut hormone (GLP-1, GIP, PYY) in fasting and post-prandial phase
Glycaemic variability | 6 months
  Change from baseline in the swings in blood glucose levels, expressed as the mean amplitude of glycaemic excursion (MAGE)
Insulin sensitivity | 6 months
  Change from baseline in the measure of insulin rise in response to blood sugar levels, expressed as the homeostasis model assessment (HOMA). HOMA estimates steady state beta cell function and insulin sensitivity as percentages of the normal reference population.
Sensory Neuropathy Testing in Prediabetic Obese Individuals | 6 months
  Change from baseline in vibration perception threshold measurement using the neurothesiometer
Douleur Neuropathique en4 Questions (DN4) | 6 months
  Change from baseline in Douleur Neuropathique en4 Questions (DN4) using seven interview questions and three physical tests.
Visual analogue score | 6 months
  Change from baseline in visual analogue score of pain, expressed as Units on a scale of 0 to 100. where 0 is worst possible health and 100 is the best possible health.
modified Total Neuropathy Score | 6 months
  Change from baseline in modified Total Neuropathy Score (mTNS) questionnaire expressed as the average of the five components
Brief Pain Inventory Short Form | 6 months
  Change from baseline in brief pain inventory short form (BPI-SF) scored as the mean of the seven interference items.

CONTACTS AND LOCATIONS:
Overall Officials: John Wilding, DM FRCP, Principal Investigator — University of Liverpool
Locations (1):
- University Hospital Aintree, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Wang Y, Ding Z, Cao G, Hu F, Sun Y, Ma Z, Zhou D, Su B. Relative validity of an indirect calorimetry device for measuring resting energy expenditure and respiratory quotient. Asia Pac J Clin Nutr. 2018;27(1):72-77. doi: 10.6133/apjcn.032017.02. PMID 29222882
- [Background] Das SK, Saltzman E, McCrory MA, Hsu LK, Shikora SA, Dolnikowski G, Kehayias JJ, Roberts SB. Energy expenditure is very high in extremely obese women. J Nutr. 2004 Jun;134(6):1412-6. doi: 10.1093/jn/134.6.1412. PMID 15173405
- [Background] Melo CM, Tirapegui J, Ribeiro SM. [Human energetic expenditure: concepts, assessment methods and relationship to obesity]. Arq Bras Endocrinol Metabol. 2008 Apr;52(3):452-64. doi: 10.1590/s0004-27302008000300005. Portuguese. PMID 18506270
- [Background] Lam YY, Ravussin E. Indirect calorimetry: an indispensable tool to understand and predict obesity. Eur J Clin Nutr. 2017 Mar;71(3):318-322. doi: 10.1038/ejcn.2016.220. Epub 2016 Nov 16. PMID 27848941
- [Background] McLay-Cooke RT, Gray AR, Jones LM, Taylor RW, Skidmore PML, Brown RC. Prediction Equations Overestimate the Energy Requirements More for Obesity-Susceptible Individuals. Nutrients. 2017 Sep 13;9(9):1012. doi: 10.3390/nu9091012. PMID 28902175
- [Background] Alves VG, da Rocha EE, Gonzalez MC, da Fonseca RB, Silva MH, Chiesa CA. Assessement of resting energy expenditure of obese patients: comparison of indirect calorimetry with formulae. Clin Nutr. 2009 Jun;28(3):299-304. doi: 10.1016/j.clnu.2009.03.011. Epub 2009 Apr 23. PMID 19398250
- [Derived] Lim J, Alam U, Cuthbertson D, Wilding J. Design of a randomised controlled trial: does indirect calorimetry energy information influence weight loss in obesity? BMJ Open. 2021 Mar 24;11(3):e044519. doi: 10.1136/bmjopen-2020-044519. PMID 33762240

DOCUMENTS (1):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT03638895/Prot_000.pdf